CLINICAL TRIAL: NCT05161624
Title: Accuracy Evaluation of Artificial Intelligence Assisted Liver Tumor Ablation Path Planning
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Huang Jinhua, Professor, Sun Yat-sen University
Other Study IDs: AIasAb
Record Dates: First submitted 2021-12-03; First posted 2021-12-17 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-12

CONDITIONS: Liver Tumor
Keywords: liver tumor; ablation; path planning; artificial intelligence; accuracy evaluation
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Path planning model
  Interventions: Diagnostic Test: Accuracy evaluation
- Junior ablation specialists
- Senior ablation specialists

INTERVENTIONS:
Diagnostic Test: Accuracy evaluation — The design of the diagnostic trial will include 160 cases of liver tumors with indications for microwave ablation after a multidisciplinary consultation with clinicians (Multiple Disciplinary Team, MDT), including primary liver cancer and metastatic liver tumors, and the tumor diameter is less than 3 cm. The test subjects consist of three groups: a. path planning model, b. junior ablation specialists, c. senior ablation specialists. The three groups will perform microwave ablation path planning on 160 selected cases of liver tumors. The attending professor of the clinical medical group of the department is responsible for scoring, evaluating whether the design of the plan is reasonable, and then comparing the scoring results by using statistical methods to evaluate the accuracy and effectiveness of the path planning model established in this study.
  Groups: Path planning model

SUMMARY:
CT-guided microwave ablation is one of the important treatment methods for primary or metastatic liver tumors. It has the advantages of minimally invasive, safe, and economical. For liver tumors with a diameter of less than 3 cm, it can be comparable to surgical resection. However, different doctors have different levels of experience, leading to a high risk of residues after ablation and even complications. The key is to fail to plan the needle placement reasonably. The past research on path planning was mostly conducted by the engineering team, so that the actual clinical needs were not considered comprehensively, and the sample size of verified cases was small, which limited the application of existing models in the clinical application. In previous study, we used artificial intelligence to segment the upper abdominal organs and construct the constraint function to establish the ablation path planning model, and initially verified the effectiveness of the path planning model in a small number of cases. Now it is planned to expand the number of patients enrolled to evaluate the accuracy of the ablation path planning model that we have established.

ELIGIBILITY:
Inclusion Criteria:

1. 18-70 years old patients with liver tumors, not limited to primary liver cancer or secondary liver metastases;
2. The number of tumors is less than 5;
3. The diameter of the tumor is less than 3 cm;
4. No local treatment of intrahepatic tumors has been done in the past.

Exclusion Criteria:

1. Diffuse liver tumor;
2. Multiple lesions in the liver> 3cm, which cannot be completely ablated;
3. Patients with lymph node metastasis and distant metastasis outside the liver;
4. Other situations where the researcher believes that it is necessary to withdraw from the study

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Liver tumor patient with goal for non-evidence disease
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2021-12-15 (Estimated); Primary Completion 2022-02-28 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
Receiver operating characteristic curve, ROC | 2 years

SECONDARY OUTCOMES:
Area under curve, AUC | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No